CLINICAL TRIAL: NCT03483181
Title: Thromboprophylaxis in Patients Undergoing Orthopedic Surgeries; Using Propensity Score Matching
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hanoi Medical University (Other)
Collaborators: Bach Mai Hospital (Other)
Responsible Party: Principal Investigator, Bui My Hanh, Director, Science Research and International Cooperation Unit, Hanoi Medical University
Other Study IDs: ĐTĐL.CN.53/16
Record Dates: First submitted 2018-03-19; First posted 2018-03-30 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Thrombosis; Deep Vein Thrombosis; Surgery--Complications
MeSH Terms: conditions — Thrombosis; Venous Thrombosis | interventions — Rivaroxaban; Enoxaparin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Orthopedic surgery patient records: Medical records from patients aged 18 years or older with orthopedic surgeries during the hospitalization
  Interventions: Drug: Xarelto (rivaroxaban); Drug: Lovenox (enoxaparin)

INTERVENTIONS:
Drug: Xarelto (rivaroxaban) — An oral anticoagulant medication for the prevention of VTE (Venous thromboembolism) related to orthopedic surgery. Patients received rivaroxaban during one day prior to or two days after orthopedic surgery during the hospitalization.
Drug: Lovenox (enoxaparin) — An injectable anticoagulant medication for the prevention of VTE (Venous thromboembolism) related to orthopedic surgery. Patients received enoxaparin during one day prior to or two days after orthopedic surgeries during the hospitalization.

SUMMARY:
Venous thromboembolism (VTE), including deep vein thrombosis (DVT) and pulmonary embolism (PE), is a common post-operative complication. The necessity for anticoagulant therapy after orthopedic surgeries is widely understood, but treatment administration patterns in the prevention of venous thromboembolism (VTE) after orthopedic surgeries during the hospital stay have yet to be examined.

The main objective of this study is to perform a comparative effectiveness review examining the benefits and harms associated with venous thromboembolism prophylaxis in patients undergoing orthopedic surgeries.

It is around efficacy and safety evaluation of using anticoagulant for thromboprophylaxis in patients undergoing orthopedic surgeries taking into the account the reliable selection of patients most benefit.

The aims of this study is to analyze patient records in teaching hospitals database of our country (including: Hanoi Medical University, Bach Mai Hospital, Cho Ray Hospital, Viet Duc University Hospital) and compare the outcomes and costs between different types of anticoagulant medications that were prescribed for the prevention of VTE following orthopedic surgeries. This analysis will assess and quantify the outcomes, resource utilization, and cost of care for patients receiving rivaroxaban or enoxaparin. The outcomes of interest include the occurence of DVT and PE, rates of major bleeds, medical resource utilization, and total costs (medical plus pharmacy).

ELIGIBILITY:
Inclusion Criteria:

* Undergo Orthopedic Surgery
* Thromboprophylaxis Decision Taken
* At least 18 years of age

Exclusion Criteria:

* Planned intermittent pneumatic compression
* A requirement for anticoagulant therapy that could not be stopped
* Severe hypersensitivity reaction (eg, anaphylaxis) to rivaroxaban or enoxaparin.
* Received another anticoagulant for more than 24 hours
* Active bleeding or a high risk of bleeding
* Thrombocytopenia associated with a positive test for antiplatelet antibody.
* Warfarin associated international normalized ratio (INR) more than 1.5 on the day of the surgery
* Conditions preventing bilateral venography
* Intensive care unit (ICU) stay after surgery
* Pregnant or breast-feeding
* Creatinine clearance less than 30 ml per minute or acute renal failure before the surgery or at any point during the study period.
* Moderate or Severe (Child Pugh B or C) hepatic Impairment or in patients with any hepatic disease associated with coagulopathy.
* Concomitant use of drugs that are both P--glycoprotein inhibitors and moderate to strong cyp3a4 (ketoconazole, itraconazole, lopinavir/ritonavir, ritonavir, indinavir/ritonavir & conivaptan)
* Creatinine clearance (CrCl) 15 to 80 mL/min and concurrent use of P-glycoprotein inhibitors or moderate CYP3A4 inhibitors (eg, abiraterone acetate, diltiazem, dronedarone, erythromycin, verapamil)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years or older who experienced a orthopedic surgeries during the hospitalization were the initial target population.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Deep-vein thrombosis (DVT) | 1 year
  The frequency of Deep-vein thrombosis
  Symptoms and signs of DVT may include unilateral leg swelling, pain in the affected leg, calf tenderness in affected leg, increased leg warmth, erythema of affected leg, or a "palpable cord" may be felt in the affected leg.
Non-fatal pulmonary embolism (PE) | 1 year
  Frequency of pulmonary embolism (non-fatal)
  Regarding Pulmonary Embolism (PE), diagnosis is suspected in patients with dyspnea, tachypnea, pleuritic chest pain, cough, and/or fever. Diagnosis begins with initial risk stratification "Wells Clinical Model for Evaluating the Pretest Probability of pulmonary embolism (PE) " based on presence of shock or persistent hypotension to identify patients at high risk of early mortality.
Mean length of hospital stay in days | 1 year
  Length of hospital stay was obtained from the discharge record and was defined as the number of days from patient admission to the hospital for orthopaedic surgeries until discharge from the hospital.
Total cost of care for index hospitalization in Vietnamese dong (VND) | 1 year
  The mean total costs (medical plus pharmacy costs) from patient records in each antithrombotic cohort from the index hospitalization
Death | 1 year
  Death from any cause including venous thromboembolism

SECONDARY OUTCOMES:
Major bleeding risk | After 4 hours of the first dose and up to 2 days after the last dose of the study drug
  The incidence of major bleeding beginning after the first dose of the study drug and up to 2 days after the last dose of the study drug (on-treatment period). Major bleeding is defined as bleeding that is fatal, occurs in a critical organ (e.g., retroperitoneal, intracranial, intraocular, and intraspinal bleeding), or requires reoperation or extra surgical-site bleeding that was clinically overt and is associated with a fall in the hemoglobin level of at least 2 g per deciliter or that requires transfusion of 2 or more units of whole blood or packed cells.
Other on-treatment bleeding | After 4 hours of the first dose and up to 2 days after the last dose of the study drug
  The incidence of major bleeding beginning after the first dose of the study drug and up to 2 days after the last dose of the study drug (on-treatment period). Major bleeding is defined as bleeding that is fatal, occurs in a critical organ (e.g., retroperitoneal, intracranial, intraocular, and intraspinal bleeding), or requires reoperation or extra surgical-site bleeding that was clinically overt and is associated with a fall in the hemoglobin level of at least 2 g per deciliter or that requires transfusion of 2 or more units of whole blood or packed cells.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code